CLINICAL TRIAL: NCT05759377
Title: Abiomed Impella V-A ECMO AUTO Mode - Observational Study
Brief Title: V-A ECMO AUTO Mode Registry
Status: Completed | Type: Observational
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-R02
Record Dates: First submitted 2023-02-22; First posted 2023-03-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: V-A ECMO AUTO Mode algorithm — The clinical effects of utilizing the V-A ECMO AUTO Mode in parallel with VA ECMO treatment shall be assessed in different clinical settings. For this, a set of relevant clinical situations and findings ("events") has been defined as trigger points where technical (via AIC) and clinical data shall be collected, linked, and analyzed. This assessment of raw data is important to further develop and adapt the software.

SUMMARY:
Abiomed Impella V-A ECMO AUTO Mode - Observational Study

DETAILED DESCRIPTION:
The overall objective of this study is to collect data during routine Impella usage in an ECpella setting to analyze and assess potential clinical effects, usability, and ease of use of an automated Impella mode to run in conjunction with a VA ECMO system for continued assessment and development of the underlying algorithms in different clinical settings.

The primary objective is thus the collection of clinical events to serve as a database for an in-silico post-hoc analysis of the V-A ECMO AUTO Mode algorithm for the Impella pump. This is accompanied by a secondary objective assessing usability, confirming the user friendliness and ease of use by collection of user experience and insights through a questionnaire and data on alarms and manual user interaction with the AIC out of the operational console data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ongoing or planned ECpella therapy

Exclusion Criteria:

* Age < 18 years
* Treatment with other than VA ECMO setup
* Treatment with Impella CP® heart pump only

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with concomitant VA ECMO and Impella CP® heart pump (ECpella) due to severe acute heart failure by any cause (e.g. cardiogenic shock in acute myocardial infarction, cardiac arrest, myocarditis).
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Gather clinical event data | Until one of the devices is permanently weaned, on average 5 days
  Collection of clinical events to serve as a database for an in-silico post-hoc analysis of the V-A ECMO AUTO Mode algorithm
Usability assessment | Until study completion, an average of 1 year
  Confirmation of usability and ease of use by collection of user data and operational console data

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kersten, MD, Principal Investigator — Uniklinik RWTH Aachen
Locations (6):
- Germany (6):
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - HDZ NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum Dresden GmbH, Dresden, Saxony
  - Universitäres Herz- und Gefäßzentrum Hamburg, Hamburg
  - UKGM Universtitätsklinikum Marburg, Marburg
  - Krankenhaus der Barmherzigen Brüder - Herzzentrum Trier, Trier

IPD SHARING:
Plan to Share IPD: No